CLINICAL TRIAL: NCT03575624
Title: Changing Health Behaviors to Manage Chronic Conditions in Community-dwelling African American Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Mary University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20170126
Record Dates: First submitted 2018-05-10; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer Female; Survivorship
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Intervention Model Description: A single arm model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition, goal-setting, yoga (Experimental): Behavioral: Nutritional and goal-setting education, yoga to promote achievement of change in health behaviors. SMART goal setting was used to guide nutritional and physical activity change to decrease disease risk and promote well-being.
  Interventions: Behavioral: Nutritional and goal-setting education, yoga

INTERVENTIONS:
Behavioral: Nutritional and goal-setting education, yoga — This integrative program series, Live Well, was delivered bi-weekly from January-May 2017, by an interdisciplinary team of a registered nurse, occupational therapist/researcher, registered dietitian, and certified yoga instructor.
  Session experiences were designed to build:
  Sisterhood for health promotion and support, Individual and group health promotion through goal-setting, Healthy family nutrition and meal planning skills , Family integrated yoga practice

SUMMARY:
The purpose of this project was to test the efficacy of partnering with a community-led wellness program to reduce disease risk and increase wellness among breast cancer survivors. Information gathered will serve the dual purpose of testing intervention effectiveness and providing the community organization data to be used to secure sustainability funding

DETAILED DESCRIPTION:
Social and environmental issues continue to impact disease morbidity and mortality resulting in the inequities of health, wellness, and quality of life experienced by African American breast cancer survivors (AABCS) living in urban Milwaukee. AABCS outcomes in Milwaukee are significantly worse (OR=1.55) than those of Caucasian survivors.

The American Diabetes Association/American Cancer Society expert committee recommends the promotion of a healthy diet, physical activity, and weight management with low waist circumference to prevent diabetes, cancer, and obesity and to extend life expectancy. According to the National Health Interview Survey, 56% of African Americans are inactive. Yoga is one way to increase physical activity while improving wellness and health in AABCS.

The investigator's goal was to facilitate improved self-care efficacy through evidence-based integrative health and wellness strategies to help families overcome the effects of multiple negative, deep-rooted social determinants.

ELIGIBILITY:
Inclusion Criteria:

* Sex: female
* Race: African American
* Survivor of breast cancer
* Physical activity participation not limited by medical doctor
* English speaking

Exclusion Criteria:

* Sex: male
* Race: not African American
* No breast cancer history
* Physical activity limitations imposed by medical doctor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change in central adiposity | 20 weeks
  circumferential measurement of waist

SECONDARY OUTCOMES:
Independent yoga posture series | 20 weeks
  participant independently demonstrates series of 6 postures
Change in body weight | 20 weeks
  weight in pounds
Change in balance | 20 weeks
  Time in seconds in single-leg stance
independent healthy meal preparation | Post intervention, after 20 weeks
  participant brings dish prepared from intervention recipe focusing on nutrition
Goal setting | 20 weeks
  Participant independently writes SMART (specific, measureable,attainable , reasonable, timely)

CONTACTS AND LOCATIONS:
Overall Officials: Julie H Hunley, PhD, Principal Investigator — Mount Mary University
Locations (1):
- Mount Mary University, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beyer KM, Zhou Y, Matthews K, Hoormann K, Bemanian A, Laud PW, Nattinger AB. Breast and Colorectal Cancer Survival Disparities in Southeastern Wisconsin. WMJ. 2016 Feb;115(1):17-21. PMID 27057575
- [Background] Garg SK, Maurer H, Reed K, Selagamsetty R. Diabetes and cancer: two diseases with obesity as a common risk factor. Diabetes Obes Metab. 2014 Feb;16(2):97-110. doi: 10.1111/dom.12124. Epub 2013 Jun 12. PMID 23668396
- [Background] NCHS, National Health Interview Survey, 2016, Sample Adult Core component retrieved online https://www.cdc.gov/nchs/data/nhis/earlyrelease/EarlyRelease201803_07.pdf
- [Background] Moadel AB, Shah C, Wylie-Rosett J, Harris MS, Patel SR, Hall CB, Sparano JA. Randomized controlled trial of yoga among a multiethnic sample of breast cancer patients: effects on quality of life. J Clin Oncol. 2007 Oct 1;25(28):4387-95. doi: 10.1200/JCO.2006.06.6027. Epub 2007 Sep 4. PMID 17785709